CLINICAL TRIAL: NCT00031096
Title: A 12-week, Randomized, Double-blind, Multicenter Study Comparing the Clinical Efficacy and Safety of Azelaic Acid 15% Gel (SH H 655 BA) With Its Vehicle (SH H 655 PBA) in Patients With Mild to Moderate Acne.
Brief Title: Comparison of Efficacy and Safety of Azelaic Acid 15% Gel With Its Vehicle in Subjects With Mild to Moderate Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90905; 304343 (90905) (Other: Company internal); 306100 (91138) (Other: Company internal); 4343 (Other: Company internal)
Record Dates: First submitted 2002-02-21; First posted 2002-02-22 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2014-02

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Propionibacterium acnes
MeSH Terms: conditions — Acne Vulgaris | interventions — azelaic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Azelaic Acid Gel 15% (Finacea, BAY39-6251)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Vehicle gel (SH H 655 PBA)

INTERVENTIONS:
Drug: Azelaic Acid Gel 15% (Finacea, BAY39-6251) — Azelaic Acid 15% gel (SH H 655 BA) applied topically two times per day.
  Arms: Arm 1
Drug: Vehicle gel (SH H 655 PBA) — Vehicle gel (SH H 655 PBA) applied topically two times per day.
  Arms: Arm 2

SUMMARY:
Comparison of efficacy and safety of Azelaic Acid 15% gel with its vehicle in male and female patients with mild to moderate acne.

Qualified subjects will apply the gel to their face twice a day for a period of 12 weeks. Subjects will be required to return to the doctor's office for up to 5 visits.

DETAILED DESCRIPTION:
Acne is a common inflammatory skin condition characterized by skin eruptions around hair follicles. People with acne can have pustules (zits or pimples), papules, whiteheads or blackheads, nodules, and redness of the skin. Acne usually involves the face and shoulders, but can also involve the chest, arms, and legs. The purpose of this study is to evaluate the safety and effectiveness of an investigational gel containing active medication compared to the same gel without any active medication (placebo or vehicle) in subjects with mild to moderate facial acne.

This study has initially been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.

Intendis Inc., a Bayer HealthCare company, is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study you MUST have:

* Predominantly facial localization of acne
* Mild to moderate acne vulgaris characterized by the presence of both inflammatory papules and/or pustules, and comedones (whiteheads/blackheads), and of a severity suitable for treatment with topical single therapy.
* a minimum of ten and a maximum of fifty inflammatory papules and/or pustules in the facial area and
* 10 to 100 comedones in the facial area
* no more than 3 small nodules (approx. 5 mm in diameter) in the facial area
* Male and female patients
* Age greater or equal to 12 years
* Ability and willingness to accept and comply with the administration of the investigational drugs over 12 weeks and to comply with the required medical examinations (signed informed consent).

Exclusion Criteria:

To be included in the study you MUST NOT have:

* Localization of acne predominantly on the chest and/or the back or confined to the chest and/or the back
* Sandpaper acne with hundreds of small facial comedones
* Moderate or severe acne requiring systemic therapy
* Multitude of small nodules and/or multiple large nodules, cysts, polyporous comedones, draining sinuses e.g. nodulocystic/conglobate acne
* Other skin conditions that might interfere with acne diagnosis and/or evaluation (such as facial psoriasis, seborrheic dermatitis, perioral dermatitis and papulopustular rosacea)
* Anticipated or scheduled hospitalization, e.g. for surgery, during the study
* Female patients who have not continuously used their present brand of oral contraceptive (if any) or other hormone therapy for at least 3 months
* Continuous concurrent use of any topical and/or systemic treatment which affects acne
* History of hypersensitivity to any ingredient of the trial drugs
* Concurrent involvement in another investigational study or participation within 30 days prior to the start of this study
* You must not have taken or have had the following types of treatment or therapy prior to being admitted into the study:

  * Oral isotretinoin (i.e. Accutane) for 6 months
  * Ortho Tri-Cyclen or Estrostep for 3 months
  * Oral antibiotics (i.e. tetracyclines, erythromycin) for 4 weeks
  * Systemic corticosteroids for 4 weeks
  * Systemic non-steroidal anti-inflammatory drugs (NSAIDs) at anti-inflammatory doses for 4 weeks
  * Topical (applied to skin) retinoid creams, ointments, gels for 2 weeks
  * Topical antibiotics (i.e. tetracyclines, erythromycin, clindamycin) for 2 weeks
  * Topical corticosteroids or topical non-steroidal anti-inflammatory (NSAIDs) drugs for 2 weeks
  * Topical imidazole antimycotics for 2 weeks
  * Topical benzoyl peroxide (BPO) for 2 weeks
  * Topical over-the-counter remedies for acne (salicylic acid) for 2 weeks If you have had any of the above, you may still qualify for the study following a washout period (time for your body to completely eliminate, or get rid of, the medication). The study doctor will evaluate whether there is anything else in your history that may affect your safety in the study or interfere with evaluations. He/she may therefore advise you not to participate.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 879 (Actual)
Dates: Start 2002-01; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
The nominal and percent change in lesions counts from baseline to last available visit (end of treatment) and treatment success rates based on Investigator's assessment of mild to moderate acne | 12 weeks

SECONDARY OUTCOMES:
Investigators rating of overall improvement and patients self assessment of overall improvement and cosmetic acceptability | 12 weeks
Adverse event reports and patient's opinion on local tolerability of the study gels at the end of study | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- United States (16):
  - Mobile, Alabama
  - Boulder, Colorado
  - Newnan, Georgia
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Albuquerque, New Mexico
  - Bay Shore, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Knoxville, Tennessee
  - Bryan, Texas
  - San Antonio, Texas
  - Seattle, Washington